CLINICAL TRIAL: NCT03230396
Title: Oral Release and Pharmacokinetics of Vitamins From a Gum-based Delivery System
Brief Title: Vitamin Gum Pharmacokinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Vitaball, Inc. (Unknown)
Responsible Party: Principal Investigator, Joshua Lambert, Associate Professor, Department of Food Science, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00001013
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Nutrient Pharmacokinetics
Keywords: vitamins; dietary supplements; chewing gum; pharmacokinetics; healthy human subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Commercially-available chewing gum not supplemented with vitamins. Contains: Sugar; Dextrose; Gum Base; Corn Syrup; Natural and artificial flavors; artificial colors; carnauba wax; resinous glaze; neotame; butylated hydroxytoluene.
  For saliva collection phase: No placebo is used. For blood collection phase: Subjects will chew two pieces at time = 0, 0.75, 4, and 8 h for 30 min at each time point.
  Interventions: Dietary Supplement: Placebo
- Vitamingum Sport (Experimental): Same gum base as placebo but supplemented with vitamins (per piece): retinyl palmitate (1250 IU); ascorbic acid (15 mg); cholecalciferol (100 IU); dl-tocopherol acetate (7.5 IU); thiamine mononitrate (375 microg); riboflavin (425 microg); niacinamide (5 mg); calcium d-panothenate (2.5 mg); pyroxidine HCl (500 microg); cyanocobalamin (1.5 microg); folic acid (100 microg); biotin (11.25 microg).
  For saliva collection phase: Subjects will chew 2 pieces for 30 min. For blood collection phase: Subjects will chew two pieces at time = 0, 0.75, 4, and 8 h for 30 min at each time point.
  Interventions: Dietary Supplement: Vitamingum Sport
- Vitamingum Immunity (Experimental): Same gum base as placebo but supplemented with vitamins (per piece): retinyl palmitate (2000 IU); ascorbic acid (62.5 mg); cholecalciferol (200 IU); dl-tocopherol acetate (20 IU); niacinamide (10 mg); calcium d-panothenate (10 mg); pyroxidine HCl (1 mg); cyanocobalamin (5 microg); folic acid (200 microg); biotin (75 microg); zinc sulfate (2.5 mg); sodium selenite (17.5 microg); chromium picolinate (60 microg); and potassium iodide (40 microg).
  For saliva collection phase: Subjects will chew 1 pieces for 30 min. For blood collection phase: Subjects will chew 1 piece at time = 0, 0.75, 4, and 8 h for 30 min at each time point.
  Interventions: Dietary Supplement: Vitamingum Immunity

INTERVENTIONS:
Dietary Supplement: Vitamingum Sport — Vitamin -supplemented chewing gum
  Arms: Vitamingum Sport
Dietary Supplement: Vitamingum Immunity — Vitamin -supplemented chewing gum
  Arms: Vitamingum Immunity
Dietary Supplement: Placebo — Control chewing gum. No vitamin content.
  Arms: Placebo

SUMMARY:
The present study will investigate the oral release and systemic pharmacokinetics of a panel water- and fat-soluble vitamins from two commercially-produced chewing gum formulations. Vitaball, Inc. (Ft. Thomas, KY) markets a line of vitamin-fortified gums. These products include Vitamingum Sport and Vitamingum Fresh, which are marketed to different consumer populations. There is currently no available data on the release of vitamins from these products in the oral cavity or the impact of chewing these products on plasma levels of the component vitamins following acute administration. The investigators hypothesize that these chewing gum products will increase both salivary and plasma levels of the component vitamins. The present study has two major objectives:

1. To determine the extent to which a subset of water-soluble and fat-soluble vitamins in two different Vitamingum products are released from the gum matrix and into the saliva as healthy human subjects chew the gum.
2. To determine the extent to which chewing Vitamingum can acutely influence plasma levels of a subset of water-soluble and fat-soluble vitamins in a population of healthy human subjects.

The test articles are commercially-marketed products and are currently available to participants outside the study (http://chewvitamingum.com). The present study is not intended to develop a treatment for a particular disease, but rather to determine if the vitamin components of these commercially-produced chewing gum products are bioaccessible or bioavailable. Vitamin supplements administered as tablets, capsules, caplets, or gummies might be regarded as the "standard of care".

DETAILED DESCRIPTION:
Study Design The study will involve two phases. The first phase will be to compare the release of the component vitamins in two chewing gum products into the saliva. This will employ a parallel design in which half the subjects (7 - 8) chew a product marketed for athletes "Sport" and half (7 - 8) chew one marketed for immune system support "Immunity". The second phase will be to compare the acute effects of chewing the two gums on plasma levels of the component vitamins. A single-blinded, double cross-over design with 15 healthy human subjects will be employed. Subjects be randomly assigned to "Sport", "Immunity", or a placebo gum matched for color and flavor but without vitamins. Each phase will be separated by a one-week washout period.

Study Procedures 1. Screening: There will be a phone screening prior to medical screening at the University Park Clinical Research Center (CRC). This will be used to establish explain the study to the prospective participant, establish eligibility and set up an appointment for the medical screen.

2 Medical Screen: Prior to acceptance into the research study, participants must complete consent forms, a medical history form, and have measurements taken (height, weight, blood pressure). If female, a urine pregnancy test will be self-administered to ensure that the subject is not pregnant. If the subject is still eligible after these tests, a small amount of blood (10 mL) will be collected by a CRC nurse using a single needle stick. The blood will be screened for markers of liver function (alanine aminotransferase, aspartate aminotransferase, or bilirubin), kidney function (blood urea nitrogen), and iron status. If a blood sample cannot be collected, the nurse try a second time, or to withdraw from the study. If a second try is unsuccessful, the participant will be excluded from the study.

3 Research Study Overview: If eligible, the subjects will have four study days (1 visit to the Food Science Building and 3 visits to the CRC). The visit to the Food Science Building will be for collection of saliva samples and will last less than 1 h. The three visits to the CRC will be to collect blood samples and will be scheduled from 7:30 am to 6:00 pm. During this day, the subject will be required to remain at the GCRC from 7:30 am to 12:30 pm. The subject will be able to leave after 6:00 pm, but will need to return at 7:30 pm for an additional blood draw.

4 Prior to Study Visits: Subjects will be required to refrain from the use of any vitamin supplement for one week prior to initiation of the study and for the duration of the study. They may consume their normal diet during the study. On the days of the "Blood Collection" visits, the subjects arrive at the CRC having not eaten breakfast. Breakfast will be provided by the investigators prior to the insertion of the catheter. The subjects should drink plenty of water on the day before and the day of the study visit.

5 Saliva Collection Visit:

a. Subjects will report to the Food Science Building at a mutually-agreed upon time.

b. Subject will be instructed to brush their teeth with a new toothbrush and toothpaste (provided by investigator) prior to the start of the session.

c. Subjects will be instructed to consume 250 mL of tap water prior to starting the chewing gum treatment.

d. Prior to chewing, an unstimulated baseline saliva sample will be collected. e. Subjects will be randomly assigned to a treatment group and given the test gum (2 pieces of gum) and instructed to chew the gum for 30 min. To standardize chewing rate, subjects will be asked to chew in time to a metronome (set to 72 beats per minute) f. Subjects will then expectorate into a centrifuge tube at 2, 5, 15, and 30 min after chewing is commenced.

g. All saliva produced during the 30 min experiment will be collected, as well the gum.

6 Blood Collection Visits:

1. The subjects will be asked to report to the CRC by 7:30 am. On each study day, the subjects will be provided with low vitamin breakfast and lunch by the investigator. The subjects will be asked to complete the meal by 8:00 am.
2. The subjects will have the option of having a numbing lotion (LMX cream containing lidocaine) applied to their arm. This anesthetic takes 30 minutes to take effect. If the subjects wish to use the lotion, they must tell the CRC study staff before the visit since it affects the experimental timing.
3. A nurse will insert an IV catheter into a vein on their arm or hand. This will allow the nurse to draw multiple blood samples without having to insert a needle each time. If the first attempt to insert the catether is unsuccessful, the nurse will make a second attempt. If a catether cannot be established, the participant will be excluded from the rest of the study. The catheter will be removed at 4:00 pm on the first day of each set of study visits. Because of the design of the research study, one additional blood sample will be collected using a separate needle insertion at 8:00 pm of the visit. This means that the subject will receive 2 needle insertions per visit.
4. Once the IV catheter is inserted, 10 mL of blood will be collected (~2 teaspoons).
5. The subject will then be asked to chew one ("immunity") or two ("sport") pieces of test gum (or 2 pieces of placebo) in time with a metronome (72 beats per min) for 30 min.
6. At 15 minutes, 30 minutes and 1.5, 4.25, and 10 hours, the nurse will collect additional 10 mL blood samples.
7. The subject will chew one ('immunity") or 2 ("sport") additional pieces of test gum (or 2 pieces of placebo) at 45 min, 4, and 8 hours after the insertion of the catheter (time 0).
8. Around noon, the subject will be given a low vitamin lunch by the CRC.
9. Because the time between blood samples increases over the course of the day, the subject will be allowed to leave the CRC following collection of the 4.25 hour 10 mL blood sample (12:30 pm). The nurse will remove the catheter at 12:30 pm. The subject will need to come back to the CRC at 6:00 pm for a 10 hour 10 mL blood collection.
10. The second and third blood draw visits will be identical to the first visit, except the subjects will be assigned to the other treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 - 60 yrs old in generally good health.
2. Healthy oral cavity with no pre-existing oral diseases including cancer, periodontitis, or mucositis.
3. No chewing or swallowing disorders.
4. No known clotting disorders.
5. Willingness to follow the investigator instructions and requirements of the protocol.
6. Ability to give consent.
7. Proficiency with the English language (both written and verbal)

Exclusion Criteria:

1. Pre-existing oral diseases including oral cancer, periodontitis, or mucositis.
2. Chewing or swallowing disorder.
3. Iron deficiency or anemia. The level of deficiency needed for exclusion will be at the discretion of the CRC physician associated with the study.
4. Pregnant, lactating, or planning to become pregnant during the study.
5. Phenylketonuric
6. Medical, social, or economic circumstance which is likely to prevent adherence to the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Salivary vitamin levels | Measured for 30 min after a single treatment with gum.
  levels of a panel of water- and fat-soluble vitamins released from gum into the saliva.
Plasma vitamin levels | Measured over the course of 10 h in a single day after chewing placebo or experimental gums.
  levels of a panel of water- and fat-soluble vitamins released from gum in blood plasma after chewing placebo or experimental gums.

IPD SHARING:
Plan to Share IPD: Yes
De-identified, aggregated saliva and blood level vitamin data, as well as de-identified individual saliva and blood vitamin levels data will be shared with other investigators upon request. We will include contact information for the study in resultant publications to allow other researchers to request the data. We will also summarize the results of the study on the PI's faculty webpage (http://foodscience.psu.edu/directory/jdl134) with contact information to request data.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available upon completion of the study and acceptance of the first manuscript describing the results of the study. It will be available for a period of 5 years.
Access Criteria: De-identified data will be made available to academic researchers and industry scientists. Requests for data will be reviewed by the study PI. Data will be supplied for research and teaching uses.

REFERENCES:
- [Background] Jacob RA, Swendseid ME, McKee RW, Fu CS, Clemens RA. Biochemical markers for assessment of niacin status in young men: urinary and blood levels of niacin metabolites. J Nutr. 1989 Apr;119(4):591-8. doi: 10.1093/jn/119.4.591. PMID 2522982
- [Background] Marszall ML, Lebiedzinska A, Czarnowski W, Makarowski R, Klos M, Szefer P. Application of the high-performance liquid chromatography method with coulometric detection for determination of vitamin B(6) in human plasma and serum. J Chromatogr B Analyt Technol Biomed Life Sci. 2009 Oct 1;877(27):3151-8. doi: 10.1016/j.jchromb.2009.08.014. Epub 2009 Aug 20. PMID 19733133
- [Background] Zhao Y, Lee MJ, Cheung C, Ju JH, Chen YK, Liu B, Hu LQ, Yang CS. Analysis of multiple metabolites of tocopherols and tocotrienols in mice and humans. J Agric Food Chem. 2010 Apr 28;58(8):4844-52. doi: 10.1021/jf904464u. PMID 20222730